CLINICAL TRIAL: NCT02444208
Title: Randomized Clinical Trial (01): A Feasibility Trial for Inhibitory-Control Training to Reduce Cocaine Use
Brief Title: A Feasibility Trial for Inhibitory-Control Training to Reduce Cocaine Use
Acronym: RCT(01)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Craig Rush, Professor, University of Kentucky
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: RCT (01); R34DA038869 (NIH)
Record Dates: First submitted 2015-05-11; First posted 2015-05-14 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Cocaine Use Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cocaine Inhibitory Control Training (Experimental): This group will receive active inhibitory control training.
  Interventions: Behavioral: Active Inhibitory Control Training
- Neutral Inhibitory Control Training (Placebo Comparator): This group will receive neutral inhibitory control training.
  Interventions: Behavioral: Neutral Inhibitory Control Training

INTERVENTIONS:
Behavioral: Active Inhibitory Control Training — Subjects will learn to inhibit responding in the presence of cocaine cues.
  Arms: Cocaine Inhibitory Control Training
Behavioral: Neutral Inhibitory Control Training — Subjects will learn to inhibit responding in the presence of neutral cues.
  Arms: Neutral Inhibitory Control Training

SUMMARY:
Cocaine abuse is an unrelenting public-health concern. Behavioral therapies are considered the "standard of care" for reducing cocaine use and preventing relapse. However, even with intense behavioral interventions, rates of relapse to cocaine use are discouragingly high (i.e., 60-95% of patients return to drug use). Novel strategies are urgently needed to improve treatment outcomes for cocaine-use disorders. The overarching goal of this project is to assess the feasibility, acceptability and initial efficacy of an innovative cocaine-based inhibitory-control training procedure. This goal will be accomplished through the conduct of a Stage I pilot trial. Cocaine-dependent participants will be enrolled and randomized to receive inhibitory-control training to cocaine or neutral images (N=20/condition). This proposed intervention, cocaine based inhibitory-control training, will be delivered using an innovative computer program which teaches cocaine abusers to inhibit a pre-potent response to cocaine or neutral cues. The primary hypothesis is the proposed procedures are feasible and acceptable to the participants. Feasibility will be assessed by determining time needed to enroll the target sample; adaptive randomization outcomes; participant attendance, completion and adherence to study procedures. Acceptability will be determined using a Treatment Acceptability Questionnaire. The secondary hypothesis is that participants receiving cocaine-based inhibitory-control training will reduce their drug use to a greater extent than their counterparts in the neutral-image condition. Reduced cocaine use will be demonstrated by fewer positive-urine samples using qualitative urinalysis and a reduction in levels of benzoylecgonine as determined by quantitative urinalysis (i.e., ELISA). The third hypothesis is that participants receiving cocaine-based inhibitory-control training will show improved inhibitory control and neurocognitive functioning relative to their counterparts in the neutral-image condition. Improved inhibitory control, impulsivity and cognitive functioning will be demonstrated using a battery of clinical instruments and laboratory tasks. The proposed research is highly innovative in that it will provide critical information regarding the feasibility, acceptability, initial efficacy of cocaine-based inhibitory-control training to reduce drug use and improve inhibitory control and neurocognitive functioning in cocaine-dependent participants. Cocaine-based inhibitory control training is also easy to administer (i.e., 15 minutes), inexpensive, need not be administered by a clinician, and could easily be incorporated into current behavioral or community-based treatment approaches to enhance sustained abstinence, thereby quickly impacting clinical research and practice.

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use verified by a cocaine-positive urine sample
* Meet Cocaine Abuse or Dependence criteria, verified by computerized Structured Clinical Interview for DSM-IV (SCID)
* Subjects must be seeking treatment for their cocaine use.
* Subjects must have at least 10% errors in response to cocaine go cues on the ABBA Task at baseline

Exclusion Criteria:

* History of serious physical or psychiatric disease that would interfere with study participation
* Current physical or psychiatric disease that would interfere with study participation
* Current or past histories of substance abuse or dependence that would interfere with study completion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Stop-Signal Task | 8 weeks after study entry
  Response inhibition and response execution will be measured using a stop-signal paradigm using a choice reaction time task that engages participants in responding to go-signals when stop-signals occasionally inform them to inhibit the response.

SECONDARY OUTCOMES:
Retention | 8, 9 and 10 weeks after study entry
  The number of subjects retained through follow up will be determined.
Recruitment | Three years
  The number of subjects recruited into the entire trial will be determined.
Treatment acceptability | 8, 9 and 10 weeks after study
  A patient treatment acceptability questionnaire will be included to determine whether patients find study procedures acceptable.
Protocol Adherence | Three years
  The number of protocol violations across the entire trial will be determined.
Self-Reported Cocaine Use | 7 days
  Self-reported cocaine use will be recorded every 7 days for 10 weeks.
Biologically verified cocaine use | 72 hours
  Cocaine use will be determined using quantitative and qualitative screens at least every 72 hours for 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Craig R. Rush, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States